CLINICAL TRIAL: NCT06078423
Title: Randomized, Blind, Phase III Clinical Trial Comparing the Immunogenicity and Safety of Freeze-dried Human Rabies Vaccine (MRC-5 Cells) With a 5-dose Program and a 4-dose (2-dose First-dose) Program
Brief Title: A Clinical Trial of Freeze-dried Human Rabies Vaccine (MRC-5 Cells)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018-Rab01
Record Dates: First submitted 2023-06-13; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Rabies Vaccine Adverse Reaction
Keywords: Safety; Efficacy

STUDY DESIGN:
Intervention Model Description: Similar vaccine control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Investigational Vaccine - 5-dose program (Experimental): Freeze-dried human rabies vaccine (MRC-5 cells), 1.0 ml after reconstitution, with a titer of not less than 5.24 IU, Anhui Zhifeilongkoma Biopharmaceutical Co., Ltd.
  Interventions: Biological: Freeze-dried human rabies vaccine (MRC-5 cells) Zhifeilongkoma - 5-dose program
- Investigational Vaccine - 4-dose program (Experimental): Freeze-dried human rabies vaccine (MRC-5 cells), 1.0 ml after reconstitution, with a titer of not less than 5.24 IU, Anhui Zhifeilongkoma Biopharmaceutical Co., Ltd.
  Interventions: Biological: Freeze-dried human rabies vaccine (MRC-5 cells) Zhifeilongkoma - 4-dose program
- Control vaccine - 5-dose program (Active Comparator): Freeze-dried human rabies vaccine (MRC-5 cells), 1.0 ml after reconstitution, with a titer of not less than 4.57 IU, ,Chengdu Kanghua Biological Products Co., Ltd
  Interventions: Biological: Freeze-dried human rabies vaccine (MRC-5 cells) Kanghua - 5-dose program
- Control vaccine - 4-dose program (Active Comparator): Freeze-dried human rabies vaccine (MRC-5 cells), 1.0 ml after reconstitution, with a titer of not less than 4.57 IU, ,Chengdu Kanghua Biological Products Co., Ltd
  Interventions: Biological: Freeze-dried human rabies vaccine (MRC-5 cells) Kanghua - 4-dose program

INTERVENTIONS:
Biological: Freeze-dried human rabies vaccine (MRC-5 cells) Zhifeilongkoma - 5-dose program — Inoculate 1 dose of Investigational vaccine each on 0, 3, 7, 14, 28 days, by intramuscular injection of deltoid muscle of upper arm
  Arms: Investigational Vaccine - 5-dose program
Biological: Freeze-dried human rabies vaccine (MRC-5 cells) Zhifeilongkoma - 4-dose program — Inoculate 1 dose of Investigational vaccine each on both arms on day 0, and 1 dose each on day 7 and 21, by intramuscular injection of deltoid muscle of upper arm
  Arms: Investigational Vaccine - 4-dose program
Biological: Freeze-dried human rabies vaccine (MRC-5 cells) Kanghua - 5-dose program — Inoculate 1 dose of Investigational vaccine each on 0, 3, 7, 14, 28 days, by intramuscular injection of deltoid muscle of upper arm
  Arms: Control vaccine - 5-dose program
Biological: Freeze-dried human rabies vaccine (MRC-5 cells) Kanghua - 4-dose program — Inoculate 1 dose of Investigational vaccine each on both arms on day 0, and 1 dose each on day 7 and 21, by intramuscular injection of deltoid muscle of upper arm
  Arms: Control vaccine - 4-dose program

SUMMARY:
This trial is a randomized, blind, similar vaccine controlled, single center, non-inferiority design phase III clinical trial, with a study population of 10 to 60 years old, conducted in two stages.Phase 1 and Phase 2

DETAILED DESCRIPTION:
This trial is a randomized, blind, similar vaccine controlled, single center, non-inferiority design phase III clinical trial, with a study population of 10 to 60 years old, conducted in two stages.

Phase 1: 40 adult subjects aged 18-60 were randomly assigned to receive the trial vaccine in a 1:1 ratio according to a 5-dose immunization program (0, 3, 7, 14, 28 days) or a 4-dose immunization program (0, 7, 21 days (2 doses for the first dose). The number of recipients for each immunization program was 20. All subjects in the adult group underwent a preliminary safety assessment 7 days after the first dose of vaccination (before the third dose of vaccine), but did not meet the suspension/termination criteria. A further 40 underage subjects aged 10-17 were enrolled in the same order as the adult group, and all subjects underwent a preliminary safety assessment 7 days after the full dose of vaccination. If they did not meet the suspension/termination criteria, they entered the second phase of the study.

Phase 2: A total of 1800 subjects aged 10 to 60 years old were randomly assigned to three groups in a 1:1:1 ratio, namely the 5-dose experimental group (vaccinated with the 5-dose program), the 5-dose control group (vaccinated with the 5-dose program), and the 4-dose experimental group (vaccinated with the 4-dose program). All subjects collected blood samples before the first dose, 7 days after the first dose, 14 days after the first dose, and 14 days after the entire dose for immunogenicity evaluation; Subjects who meet the requirements for immune persistence observation in the plan shall collect blood samples 3 months after the full vaccination, and the experimental group subjects shall also collect blood samples 12 months after the full vaccination for immune persistence evaluation.

Collect all AEs from participants within 30 minutes after each dose, collected AEs within 0-7 days after each dose (if the interval from the current dose to the next dose is less than 7 days, the collection period shall be based on the actual interval between the two doses), all non collected AEs within 30 days after the first dose to the entire dose, and all serious adverse events (SAE) within 6 months after the first dose to the entire dose.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 10 to 60 years old;
* Willing to participate in this experiment and sign an informed consent or notification form;
* The subjects themselves or/and their guardians promise to comply with the requirements of the clinical research protocol;
* Under the age of 14 (including 14 years old), the axillary body temperature is less than 37.5 ℃, and above the age of 14, the axillary body temperature is less than 37.3 ℃

Exclusion Criteria:

* Have a history of rabies vaccine immunization or use of rabies virus passive immunity preparations;
* Have a history of injury to dogs or other mammals within 12 months prior to the first vaccination;
* Have used blood products within 4 months before the first vaccination;
* Inoculate any vaccine within 14 days before the first vaccination;
* Have used other research or unregistered products (drugs or vaccines) within one month before the first vaccination, or have planned to participate in other clinical studies after enrollment in this clinical study;
* Suffering from congenital or acquired immune deficiency. Receiving immunosuppressive therapy, such as long-term (oral) systemic glucocorticoid therapy (continuous (oral) systemic glucocorticoid therapy for more than 2 weeks, such as prednisone or similar drugs);
* Have a history of convulsion, epilepsy, encephalopathy, psychosis or family history;
* Allergic to any component in the study vaccine (such as human albumin, disodium hydrogen phosphate, sodium dihydrogen phosphate, sodium chloride, sucrose, maltose, etc.); Have a history of severe allergies, such as allergic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, and local allergic necrosis reaction (Arthur reaction);
* Have any previous history of serious side effects from vaccines or drugs, such as urticaria, skin eczema, respiratory difficulties, vascular and neurological edema, etc;
* Individuals with acute febrile diseases (body temperature ≥ 38.5 ℃) and infectious diseases within 3 days before vaccination;
* Having congenital heart disease, developmental disorder or chronic disease, such as asthma, diabetes, thyroid disease;
* Suffering from urticaria within one year before receiving the experimental vaccine;
* Blood pressure: systolic blood pressure ≥ 160mmHg or diastolic blood pressure ≥ 100mmHg (regardless of medication);
* Suffering from thrombocytopenia or other coagulation disorders (which may cause contraindications for intramuscular injection);
* Women of childbearing age who have a positive urine pregnancy test, or have a fertility plan during pregnancy, lactation, or within 2 months;
* Any situation that the researcher believes may affect the evaluation of the experiment

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1880 (Actual)
Dates: Start 2019-10-19 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Antibody positive conversion rate - Immunogenicity endpoint | up to 14 days after the first/full dose of vaccination
  Antibody positivity conversion rates in the 4-dose experimental group, 5-dose experimental group, and 5-dose control group
Geometric mean concentration - Immunogenicity endpoint | 14 days after the first/full dose of vaccination
  GMC of the 4-dose experimental group, 5-dose experimental group, and 5-dose control group
Incidence of Adverse Events [Safety and Tolerability] | within 30 minutes after each dose of vaccination
  The incidence of any local and systemic adverse events (AEs)
Incidence of Adverse Events [Safety and Tolerability] | within 0-7 days after each dose of vaccination
  The incidence of collected AEs
Incidence of Adverse Events [Safety and Tolerability] | within 30 days after the first dose of vaccination to the full course of vaccination
  The incidence of non solicited AE
Incidence of Adverse Events [Safety and Tolerability] | within 6 months after the first dose administration and the entire vaccination process
  The incidence of all serious adverse events (SAE)

SECONDARY OUTCOMES:
Antibody positive conversion rate - Immunogenicity endpoint | 7 days after the first dose of vaccination；3 month after full dose of vaccination；
  Antibody positivity conversion rates in the 4-dose experimental group, 5-dose experimental group, and 5-dose control group
Geometric mean concentration - Immunogenicity endpoint | 7 days after the first dose of vaccination;3 month after full dose of vaccination；
  GMC of the 4-dose experimental group, 5-dose experimental group, and 5-dose control group
Antibody positive conversion rate - Immunogenicity endpoint | 12 month after full dose of vaccination；
  Antibody positivity in the 5-dose and 4-dose test groups
Geometric mean concentration - Immunogenicity endpoint | 12 month after full dose of vaccination；
  GMC of the 5-dose and 4-dose test groups

CONTACTS AND LOCATIONS:
Overall Officials: Fangjun Li, Bachelor, Principal Investigator — Hunan Provincial Center for Disease Control and Prevention
Locations (1):
- Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No